CLINICAL TRIAL: NCT03293810
Title: Glybera Registry, Long-term Safety and Efficacy Follow-up in Lipoprotein Lipase Deficient (LPLD) Patients Treated With Alipogene Tiparvovec (GLYBERA®)
Brief Title: Glybera Registry, Lipoprotein Lipase Deficient (LPLD) Patients
Acronym: GENIALL
Status: Completed | Type: Observational
Sponsor: UniQure Biopharma B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: REG-uQ-Glyb-001
Record Dates: First submitted 2015-05-20; First posted 2017-09-26 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Lipoprotein Lipase Deficiency; Familial Hyperlipoproteinemia Type 1; Familial Hyperchylomicronemia
MeSH Terms: conditions — Hyperlipoproteinemia Type I | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observational study — Post-Authorization Safety Study

SUMMARY:
Lipoprotein lipase deficiency (LPLD) is a rare autosomal recessive disorder, characterized by loss-of function mutations in the LPL gene, leading to the inability to produce functionally active lipoprotein lipase (LPL). LPL is the key enzyme in the metabolism of triglyceride (TG)-rich lipoproteins (chylomicrons (CM) and very low-density lipoproteins (VLDL)). LPLD results in extremely high concentrations of circulating TG-rich lipoproteins.

No drug therapy for LPLD is currently available. Clinical management of LPLD patients consists of severe dietary fat restriction and the use of medium-chain triglycerides to substitute for normal dietary fats.

Alipogene tiparvovec (Glybera®) received marketing authorisation from the European commission on 25 October 2012. Glybera® aims to correct lipoprotein lipase deficiency sufficiently to decrease the morbidity and lower the risk of inherent complications of LPLD, in adult patients genetically diagnosed with LPLD.

The Glybera Registry is designed to collect the long-term safety and efficacy data of GLYBERA®

DETAILED DESCRIPTION:
All patients treated with GLYBERA®, in a clinical trial and when GLYBERA® was commercially available who are currently participating in the LPLD Registry (Long term follow up of safety and efficacy in LPLD), will be asked to continue their participation in this Glybera Registry to collect long-term safety and efficacy data.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with GLYBERA®, either during their participation in a clinical trial or in the commercial setting till October 25th, 2017 (= expiration date of Marketing Authorization of GLYBERA®), and
* Who are currently participating in the LPLD Registry

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with GLYBERA®, either during their participation in a clinical trial or in the commercial setting till October 25th, 2017
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2014-06-27 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Long-term collection of Safety and Efficacy of GLYBERA®, as measured by collection of Adverse Events, Immunological responses and information on Pancreatitis-events | 15 years
  Adverse Events will be collected as reported by the patients during routine visits/contacts.
  Immunological responses defined as antibody formation and T-cell responses against the AAV1-capsid and against the LPLS447X transgene product, measured just before dosing and at 6 and 12 months post-dosing.
  Pancreatitis-events will be collected as reported by the patients during routine visits/contacts

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Averna, Prof, Study Chair — Universitaria Policlinico Paolo Giaccone, Palermo
Locations (1):
- Interdisciplinary Metabolism Center, Lipid Out-Patient-Clinic, Lipid Apheresis, Charité, University of Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided